CLINICAL TRIAL: NCT03726827
Title: Screening for Undiagnosed NAFLD and NASH
Brief Title: A Self Selected Population Study of Undiagnosed NAFLD and NASH, Using an Echosens FibroScan, in at Risk Populations
Acronym: SUNN
Status: Completed | Type: Observational
Sponsor: Fatty liver Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: flf-screen 1
Record Dates: First submitted 2018-10-17; First posted 2018-11-01 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: NAFLD; NASH - Nonalcoholic Steatohepatitis; Cirrhosis, Liver; Fatty Liver
Keywords: NAFLD; NASH; cirrhosis; fatty liver; incidence; fibroscan
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis; Fatty Liver; Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- population: self selected members of the general population who perceive a value in having a Fibroscan screening test of their liver
  Interventions: Other: Fibroscan screening

INTERVENTIONS:
Other: Fibroscan screening — A single Fibroscan screening for fat content and liver stiffness

SUMMARY:
Liver disease (NAFLD) and (NASH) are a rapidly increasing population health threat driven primarily by diet and lifestyle. Fibrotic liver disease, culminating in cirrhosis, is frequently asymptomatic so it is common for a patient to first learn of what is a life threatening condition by being told that they have cirrhosis. Management and treatment of cirrhosis is complex and very costly with the only current cure being a very expensive transplant for end stage liver disease. The SUNN study seeks to perform Fibroscan wellness testing on at risk but asymptomatic self selected patients in the general population to identify disease early and to triage patients toward care or educational tools based upon test results. No personally identifiable information will be collected but demographic and test results will be imported into a registry for data analysis. Results of the study will guide development of screening protocols to identify early stage disease in a wellness screening model.

DETAILED DESCRIPTION:
The standard of care published by the American Association for the Study of Liver Disease, (AASLD) do not recommend screening of asymptomatic patients for liver fibrosis so it is common that the first a patient learns of the disease is when they are diagnosed with cirrhosis. Detection at early stages of the disease process is mostly accidental as a result of other procedures.

Research has clearly established the health risks associated with liver disease and comorbidity with a wide range of other illnesses. FibroScan has been shown to be a useful test to identify asymptomatic liver disease.

The FibroScan device (Echosens) works by measuring shear wave velocity. In this technique, a 50 megahertz wave is passed into the liver from a small transducer on the end of an ultrasound probe. The probe also has a transducer on the end that can measure the velocity of the shear wave (in meters per second) as this wave passes through the liver. The shear wave velocity can then be converted into liver stiffness, which is expressed in kilopascals. Essentially, the technology measures the velocity of the sound wave passing through the liver and then converts that measurement into a liver stiffness measurement; the entire process is often referred to as liver ultrasonographic elastography. The procedure is non-invasive and presents no bio-chemical hazards as it uses only well understood ultrasound technology.

The goal of this screening study is to gather FibroScan data from the at-risk but undiagnosed population on a self-selection basis so that incidence rates can be calculated and the economics of a single function screening service can be evaluated.

The objective is to develop evidence based information to determine if noninvasive screening of at risk, comorbid people is feasible with this modality.

Furthermore, a secondary goal is to educate all participants about liver disease, lifestyle, healthy diets, organ donation, and clinical trials as part of the Foundation's larger mission of being patient advocates.

Questions Posed by this Study:

* What population demographics justify routine screening on a cost benefit basis?
* What operating cost burden is required to sustain a mobile screening project and what is the minimum utilization required to justify it?
* What portion of the asymptomatic patient with advanced disease will be willing to learn about clinical trials?

All patients will receive education about liver disease as part of the intake process. From the patient perspective, the key result will be that they receive the printed output from their FibroScan test. Interpretation of that result requires expert support. The investigators will direct patients to local medical resources where their questions can be answered, but the ideal route will be a triage through telemedicine with a hepatologist as a way to quickly direct them to proper resources. Patients with test results indicating no active disease will be offered connections to nutrition and dietary support. In all cases patients will be offered enrollment in online educational tools.

ELIGIBILITY:
Inclusion Criteria:

* self selected

Exclusion Criteria:

* Must be over 17 years old
* Cannot be pregnant
* Cannot have any implanted electronic devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General population on a self selected basis, however, recruitment efforts will be directed to the high risk population that is over 50 years old, obese, type 2 diabetic, or have other common co-morbid conditions
Sampling Method: Probability Sample
Enrollment: 1006 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Calculate the frequency distribution and severity of steatosis stage (S0, S1, S2, S3) and liver fibrosis stage (F0, F1, F2, F3, F4) in the test population. | The test period will be six months and results will be reported 3 months after end of testing.
  The frequency distribution is the percentage each stage represents of the total. Severity is described by the disease staging. Staging is not measured directly so test scores are normalized to a stage using cutoff values. The results are fat content (steatosis) and liver fibrosis (steatohepatitis) derived from test measurements of CAP score (controlled attenuation parameter) and LSM (liver stiffness measure). These are used to calculate the frequency distribution and staging of steatosis stage (S0, S1, S2, S3) and liver fibrosis stage (F0, F1, F2, F3, F4). The resulting dataset will then be assigned to a disease stage according to the breakpoints below.
  CAP S0 (<225) S1 (225-275), S2 (276-300), S3 (>300)
  LSM F0 (<7.0) F1 (7.0-7.4) F2 (7.5-9.9) F3 (10.0-13.9) F4 (>13.9)
  The distribution of the normalized dataset will be calculated as the percentage each bracket is of the total number of tests in that subset.

SECONDARY OUTCOMES:
Calculate the frequency distribution and severity of steatosis and liver fibrosis in the test population by ethnicity. | The test period will be six months and results will be reported 3 months after end of testing.
  Repeat the analysis by ethnicity

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Eskridge, BS, Principal Investigator — Fatty liver Foundation
Locations (1):
- Fatty Liver Foundation, Texas City, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
No personally identifiable information will be collected but the population data will be made available to other researchers though the method has not yet been determined

DOCUMENTS (2):
  • Informed Consent Form (2018-10-05): https://cdn.clinicaltrials.gov/large-docs/27/NCT03726827/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-10-05): https://cdn.clinicaltrials.gov/large-docs/27/NCT03726827/Prot_SAP_001.pdf